CLINICAL TRIAL: NCT00319371
Title: Registration of Skin-Temperatures and Sleep-Wake Behaviour in the Daily Life of Women With Vasospasm in Comparison to Controls
Brief Title: Registration of Skin-Temperatures and Sleep-Wake Behaviour
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Selim Orgül, MD, University Hospital, Basel, Switzerland
Other Study IDs: 074-GOB-2006-001; 02/06
Record Dates: First submitted 2006-04-04; First posted 2006-04-27 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Vasospastic Syndrome
Keywords: vasospasm; circadian; sleep-disorders
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: women with vasospasm and difficulties of initiating sleep
- 2: women without vasospasm and no difficulties of initiating sleep

SUMMARY:
We study the skin-temperature (skin temperature measurement on different skin regions) and circadian rest-activity cycles (wrist activity monitoring) of 40 women in their daily life.

This project will provide further information at which circadian phase vasospasms occur in daily routine life (one week recordings). Special interest lays on the time before sleep. The attained results could be used to establish a therapy with few side effects for people with difficulties initiating sleep because of vasospasm.

DETAILED DESCRIPTION:
We study the skin-temperature and circadian rest-activity cycles of 40 women in their daily life.

20 women with vasospasm and difficulties of initiating sleep and 20 women without vasospasm and no difficulties of initiating sleep.

Women without contraceptives will be examined in the luteal phase (i.e. in the two weeks before menstruation). The ambulant registry will be done continuously during one week with so called i-Buttons (IButtonTM, Maxim, USA). These will be fixed to various parts of the body (i.e. wrist, ankle, …) with Fixomull, a medical bond. Also the subjects have to wear a instrument for registration activity, the so called Actiwatch (Cambridge, UK). The data that will be gained from these instruments, shall help us to objectify sleep-latency and sleep-fragmentation ("sleeping-through").

Furthermore, the subjects obtain a sleep-and activity-dairy, that has to be filled before and after sleeping. At one day, that the proband can choose, saliva samples have to be taken by the subjects themselves. In the saliva, the concentration of melatonin will be qualified. The attained results could be used to establish a therapy with few side effects for people with difficulties of initiating sleep because of vasospasm.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have to show a vasospasm and difficulties of initiating sleep (screening with questionnaires and interview)
* Controls have to show no vasospasm and no difficulties of initiating sleep (screening with questionnaires and interview)

Exclusion Criteria:

* bad health or unhealthy conditions
* allergies (i.e. nickel)
* medication
* BMI<18
* migraine
* delayed sleep phase syndrome
* advanced sleep phase syndrome
* alcohol- or drug problems
* smokers
* blood donation in last three months before study
* participation at an other clinical study in last three months before study
* shift work in last three months before study
* long-distance flight (> 2 time zones) in last month before study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women with vasospasm and difficulties of initiating sleep and women without vasospasm and no difficulties of initiating sleep
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2005-11; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Eye Clinic Basel
Locations (1):
- University Eye Clinic Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- See also: Related Info — http://www.kantonsspital-basel.ch
- See also: Related Info — http://www.chronobiology.ch